CLINICAL TRIAL: NCT00817973
Title: Differential Effects of Protein Quality on Postprandial Lipemia in Response to a Fat-Rich Meal in Type 2 Diabetes: Comparison of Whey, Casein, Gluten, and Cod Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Obesity Research Centre (Other); Nordic Centre of Excellence (Other)
Responsible Party: Kjeld Hermansen, Professor, Chief Physician, MD, Dr.Med.Sci, Department of Endocrinology and Metabolism, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-PPL (5A) LSM
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes; Postprandial Lipemia
Keywords: Whey protein; gluten; casein; cod protein; GLP-1; postprandial; triglyceride; free fatty acids; chylomicrons; retinyl palmitate; type 2 diabetes; GIP; Postprandial incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caseins; Whey; CVD protocol; Glutens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Casein (Active Comparator)
  Interventions: Dietary Supplement: Casein
- Whey (Active Comparator)
  Interventions: Dietary Supplement: Whey
- Cod (Active Comparator)
  Interventions: Dietary Supplement: Cod
- Gluten (Active Comparator)
  Interventions: Dietary Supplement: Gluten

INTERVENTIONS:
Dietary Supplement: Casein
  Arms: Casein
Dietary Supplement: Whey
  Arms: Whey
Dietary Supplement: Cod
  Arms: Cod
Dietary Supplement: Gluten
  Arms: Gluten

SUMMARY:
Enhanced and prolonged postprandial triglyceride responses involve increased cardiovascular risk in type 2 diabetes. It has been demonstrated that dietary fat and carbohydrates profoundly influence postprandial hypertriglyceridemia in type 2 diabetes, whereas little information exists about the effect of proteins.

The purpose of this study is to compare the effects of the proteins casein, whey, cod, and gluten on postprandial lipid and incretin responses to a high-fat meal in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes

Exclusion Criteria:

* Liver, Kidney- and/or Heart Disease
* Serious Hypertension (160/110 mmHg)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)

PRIMARY OUTCOMES:
Triglyceride levels | 0h- 2h- 4h- 6h- 7h- 8h postprandial

SECONDARY OUTCOMES:
Incretin levels | 0h- 0.5h- 1h- 2h- 4h- 6h- 8h postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Professor, MD, Principal Investigator — Department of Endocrinology and Metabolism
Locations (1):
- Department of Clinical Nutrition, Aarhus, Denmark

REFERENCES:
- [Derived] Mortensen LS, Thomsen C, Hermansen K. Effects of different protein sources on plasminogen inhibitor-1 and factor VII coagulant activity added to a fat-rich meal in type 2 diabetes. Rev Diabet Stud. 2010 Fall;7(3):233-40. doi: 10.1900/RDS.2010.7.233. Epub 2010 Nov 10. PMID 21409315
- [Derived] Mortensen LS, Hartvigsen ML, Brader LJ, Astrup A, Schrezenmeir J, Holst JJ, Thomsen C, Hermansen K. Differential effects of protein quality on postprandial lipemia in response to a fat-rich meal in type 2 diabetes: comparison of whey, casein, gluten, and cod protein. Am J Clin Nutr. 2009 Jul;90(1):41-8. doi: 10.3945/ajcn.2008.27281. Epub 2009 May 20. PMID 19458012